CLINICAL TRIAL: NCT07296666
Title: Adjuvant Therapy for Stage II/III Cholangiocarcinoma Based on 3D-PTA Susceptibility Testing: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Adjuvant Chemotherapy for BTC Based on 3D-PTA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GWK-2025-008
Record Dates: First submitted 2025-11-24; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Cholangiocarcinoma
Keywords: BTC
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Drug Therapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group: Capecitabine + 3D-PTA-selected chemotherapy drugs (conventional dosage) (Experimental)
  Interventions: Drug: Chemotherapy (preferably with a single chemotherapeutic agent) combined with capecitabine (including capecitabine monotherapy: when the preferred drug identified is capecitabine alone).
- Control group: Capecitabine (Active Comparator)
  Interventions: Drug: capecitabine alone as adjuvant treatment

INTERVENTIONS:
Drug: Chemotherapy (preferably with a single chemotherapeutic agent) combined with capecitabine (including capecitabine monotherapy: when the preferred drug identified is capecitabine alone). — Chemotherapy combined with capecitabine (including capecitabine monotherapy) guided by 3D-PTA drug sensitivity testing versus capecitabine alone as adjuvant treatment.
  Arms: Treatment group: Capecitabine + 3D-PTA-selected chemotherapy drugs (conventional dosage)
Drug: capecitabine alone as adjuvant treatment — capecitabine alone as adjuvant treatment
  Arms: Control group: Capecitabine

SUMMARY:
This is a prospective, open-label, controlled, multicenter clinical study designed to observe and evaluate the efficacy and safety of chemotherapy (including capecitabine monotherapy) guided by 3D-PTA drug sensitivity testing versus capecitabine monotherapy as adjuvant treatment in patients with stage II/III cholangiocarcinoma after surgery.

DETAILED DESCRIPTION:
All participants underwent baseline disease assessment, including radiological evaluation within 14 days before treatment initiation. The study compared capecitabine combined with 3D-PTA-selected chemotherapy drugs (administered at standard doses) versus capecitabine monotherapy. Participants received study drugs on Day 1 of each cycle for 8 cycles. Tumor efficacy evaluation, vital signs, ECOG performance status (PS) score, physical examination, and quality of life (QoL) assessments were conducted every 9 weeks after the first dose until disease progression, unacceptable toxicity, or participant withdrawal. Adverse event (AE) monitoring and concomitant medication documentation were performed continuously from treatment initiation through 30 days post-treatment. Follow-up included tumor efficacy evaluation and QoL assessment every 6 months, with survival follow-up for participants experiencing disease recurrence or metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of written informed consent prior to participation;
2. Age ≥18 years, regardless of sex;
3. Histologically confirmed stage II/III biliary tract malignancies (including intrahepatic cholangiocarcinoma, extrahepatic/hilar cholangiocarcinoma, gallbladder cancer, distal bile duct cancer, or ampullary cancer);
4. Must have undergone radical resection (R0/R1), including liver/pancreatic resection or, less commonly, both;
5. ECOG performance status (PS) score: 0-1;
6. Expected survival >6 months and ability to tolerate combined therapy;
7. Adequate organ function (without blood component or growth factor support within 14 days):
8. Hematology: Neutrophils ≥1,500/mm³, platelets ≥100,000/mm³, hemoglobin ≥9 g/dL;
9. Liver/kidney function: Serum creatinine (SCr) ≤1.5×ULN or creatinine clearance ≥50 mL/min (Cockcroft-Gault formula); total bilirubin (TBIL) ≤2×ULN; AST/ALT ≤3×ULN; urine protein <2+ (if ≥2+, 24-hour urine protein ≤1 g); Biliary drainage: Adequate surgical drainage, no signs of infection;
10. Normal coagulation function, no active bleeding or thrombotic disease:INR ≤1.5×ULN, APTT ≤1.5×ULN, PT ≤1.5×ULN;
11. Contraception:

    1. Non-surgically sterilized or reproductive-age patients must use medically approved contraception (e.g., IUD, oral contraceptives, condoms) during and for 3 months after treatment;
    2. Reproductive-age females must have negative serum/urine pregnancy test (HCG) within 7 days before enrollment and must not be breastfeeding;
    3. Reproductive-age males must agree to use contraception with partners during and for 3 months after treatment;
12. Voluntary participation, good compliance, and willingness to follow up for safety and survival assessments.

Exclusion Criteria:

1. Early-stage BTC patients;
2. Pancreatic cancer patients;
3. Patients who have undergone other postoperative radiotherapy/chemotherapy; preoperative chemoradiotherapy followed by radical resection, but postoperative pathology still indicates Stage II/III disease is allowed;
4. Incomplete surgical recovery or unresolved biliary obstruction;
5. Patients with radiologically confirmed distant metastasis;
6. Patients with a history of or concurrent other malignancies (except for cured basal cell carcinoma of the skin and in-situ carcinoma of other sites);
7. Known allergies to any component of the investigational drug;
8. Factors significantly affecting oral drug absorption, such as inability to swallow, chronic diarrhea, or intestinal obstruction;
9. Patients with any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, or hypothyroidism; patients with vitiligo or childhood asthma that has been completely resolved and requires no intervention in adulthood may be included; patients requiring bronchodilators for medical intervention due to asthma cannot be included);
10. Patients using immunosuppressants or systemic/absorbable local corticosteroids for immunosuppressive purposes (dose >10 mg/day prednisone or equivalent) and continuing use within 2 weeks prior to enrollment;
11. Symptomatic ascites or pleural effusion requiring therapeutic paracentesis or drainage;
12. Poorly controlled cardiac symptoms or diseases, such as:

    1. NYHA Class II or higher heart failure,
    2. unstable angina,
    3. myocardial infarction within 1 year,
    4. clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
13. Coagulation abnormalities (PT >16s, APTT >43s, TT >21s, Fbg >2g/L), bleeding tendency, or receiving thrombolytic/anticoagulant therapy;
14. Active infection or unexplained fever >38.5°C during screening or before the first dose;
15. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks before the first dose;
16. History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, or severe lung dysfunction;
17. Congenital or acquired immunodeficiency, such as HIV infection, or active hepatitis (liver enzymes not meeting inclusion criteria; for hepatitis B: HBV DNA ≥103/ml; for hepatitis C: HCV RNA ≥103/ml); chronic HBV carriers with HBV DNA <2000 IU/ml (<104 copies/ml) may be included if receiving antiviral therapy during the trial;
18. Participation in other drug-related clinical trials within 1 month before enrollment or potential receipt of other systemic anti-cancer therapies during the study;
19. Live vaccination within 4 weeks before the first dose or planned during the study;
20. History of substance abuse, alcoholism, or drug addiction;
21. Inability or unwillingness to bear the cost of self-funded examinations and treatments;
22. Other factors deemed by the investigator to exclude the patient, such as severe diseases (including mental illness) requiring treatment, significant laboratory abnormalities, or family/social factors that may compromise patient safety or data/sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
12-month PFS rate. | 12-month
  12-month PFS rate.

SECONDARY OUTCOMES:
median Recurrence-Free Survival（mRFS） | 12-month
  mRFS
median Overall Survival（mOS） | 12-month
  mOS

CONTACTS AND LOCATIONS:
Overall Officials: Lu Wang, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No